CLINICAL TRIAL: NCT05302934
Title: Prospective, Multinational Pilot Study for Evaluation of the PHENO4U Data Platform in Total Knee Arthroplasty Patients
Brief Title: Evaluation of the PHENO4U Data Platform in Patients Undergoing Total Knee Arthroplasty
Acronym: Pheno4U Pilot
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2113
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Osteoarthritis; Rheumatoid Arthritis; Posttraumatic Arthropathy; Chronic Instability of Knee; Stiffness of Knee; Deformity Knee
Keywords: bi-condylar knee replacement; severe knee joint conditions; patient reported outcome
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pheno4U: The study will collect data for each patient receiving an Aesculap TKA implant. The data set will be analyzed for critical risk factors among implant and patient data in order to optimize patient-centered therapies.
  Interventions: Device: Pheno4U

INTERVENTIONS:
Device: Pheno4U — Total Knee Arthroplasty represents a well-established, reliable and successful treatment option for end-stage bicompartmental osteoarthritis or other indications resulting in joint destruction. In general, Implantation of a total knee prosthesis improves the quality of life through pain alleviation, deformity correction, joint stabilization, and/or functional range of motion (ROM) through restoration of normal knee kinematics and functionality
  Other Names: Total Knee Arthroplasty

SUMMARY:
Prospective, multinational pilot study for evaluation of the Pheno4U data platform in Total Knee Arthroplasty (TKA) patients

DETAILED DESCRIPTION:
The study will collect data for each patient receiving an Aesculap Total Knee Arthroplasty (TKA) implant. The data set will be analyzed for critical risk factors among implant and patient data in order to optimize patient-centered therapies.

The products under investigation will be used in routine clinical practice and according to the Instructions for Use (IFU). Data obtained in routine clinical use will be collected in the Pheno4U data platform. In addition, patients are expected to answer questionnaires about their health status. Furthermore, patients are asked to use the so called "BPMpathway" sensor and application in order to measure the active Range of Motion (ROM). The sensor can also be used for pre- and postoperative training .

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a total knee arthroplasty with a B. Braun knee implant system
* Signed written informed consent
* Patient's willingness & ability to use the "BPMpathway"sensor
* Patient's willingness & ability to use the "4Patient" application

Exclusion Criteria:

* Patient age < 18 years
* Patient not willing to participate at the further follow-up
* Pregnancy
* If intraoperatively an implant from a different manufacturer is used, the study patient has to be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively. No selection besides the inclusion and exclusion criteria will take place. Four different TKA implant systems can be used within the study: Columbus, E.motion, Enduro and VEGA according to the instructions for use.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Identification of any unknown risks or side effects in Total Knee Arthroplasty by using sensors and patient apps | up to 12 months postoperatively
  The study will collect data for each patient receiving an Aesculap TKA implant. The data set will be analyzed for critical risk factors among implant and patient data in order to optimize patient-centered therapies

SECONDARY OUTCOMES:
Change of Knee Injury and Osteoarthritis Outcome score | 2 weeks prior to surgery, 6 weeks postoperatively and approximately 1 year after surgery
  The Patient self-assessed Injury and Knee Osteoarthritis Outcome Scores (KOOS) is a joint-specific instrument: The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change of Hospital for Special Surgery (HSS) Knee Surgery Expectations Survey | 2 weeks prior to surgery, 6 weeks postoperatively and approximately 1 year after surgery
  The Hospital for Special Surgery (HSS) Knee Surgery Expectations Survey is a 17 item questionnaire. The survey is comprised of five different categories of expectations: pain, walking, psychological state, essential activities and non-essential activities. The responses range from ''very important'' (score: 1) to ''this does not imply to me'' (score: 5). The total summed raw score ranges from 0 to 76 and the transformed score [ = (raw score/76)×100] ranges from 0 to 100. Higher scores indicate expecting more improvement for more items.
Change of Pain | 2 weeks prior to surgery, 6 weeks postoperatively and approximately 1 year after surgery
  Information on pain is collected by the so called "painDETECT" questionnaire, a self-reported screening tool for the identification of neuropathic pain. The questionnaire contains seven weighted sensory descriptors, one item relating to spatial pain characteristics and one item relating to temporal characteristics. A total score ranging from -1 to 38 can be calculated. The total score is divided into three categories (unlikely neuropathic pain (<13), unclear (13-18), likely neuropathic pain (>18)).
Patient satisfaction | approximately 9 months after surgery
  Based on a single question 9 months after surgery patients are asked to grade their level of satisfaction with the methodology and rehabilitation procedure. They can choose between "very dissatisfied", "dissatisfied", "satisfied" or "very satisfied".
Net Promoter Score | approximately 12 months after surgery
  The Net Promoter Score (NPS) is an index ranging from -100 to 100 that measures the willingness of patients to recommend the treatment to others. It is used as a proxy for gauging the patient's overall satisfaction with a treatment. Patients are surveyed on one single question. They are asked to rate on an 11-point scale the likelihood of recommending the treatment to a friend or colleague. "On a scale of 0 to 10, how likely are you to recommend the same treatment to a friend or a colleague?" Based on their rating, customers are then classified in 3 categories: detractors, passives and promoters. 'Detractors' gave a score lower or equal to 6. 'Passives' gave a score of 7 or 8. 'Promoters' answered 9 or 10. The NPS is determined by subtracting the percentage of customers who are detractors from the percentage who are promoters.
Change of Depression, Anxiety and Stress Scale - 21 Items | 1 week prior to surgery and 2 weeks postoperatively
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items with a four point rating scale (ranging 0 - 3 points) for each item. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. The total score is calculated by summing the scores for the relevant items, the minimum score is 0 points, the maximum score for each section is 21. A lower score represents less depression, anxiety and stress.
Development of Active Range of Motion | up to 3 months after surgery
  The active Range of Motion (ROM) is measured with the BPMpathway sensor and application 3 times per day for the entire duration of usage of the sensor. In general, the sensor is used for pre- and postoperative training. Patients are expected to use the sensor from pre-op consultation up to 3 month after surgery.

OTHER OUTCOMES:
Cumulative Radiological Evaluation | for each x-ray taken in clinical routine up to last follow-up approximately 12 months postoperatively
  Imaging will be used to evaluate the implant status as well as device condition and potential presence of device-related Adverse Events including fracture, wear, loosening or radiolucencies.
Cumulative Rate of (Serious) Adverse Events | up to last follow-up approximately 12 months postoperatively
  During the course of the study any upcoming intra- or postoperative (serious) adverse events directly or possibly related to the products under investigation will be documented in the dedicated electronic case report forms (eCRFs). Recorded complications will be categorized and analyzed in order to assess the safety of the investigational products.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, Prof. Dr., Principal Investigator — Universitätsklinikum Carl Gustav Carus
Locations (4):
- Germany (3):
  - Vincentius Krankenhaus, Konstanz, Baden-Wurttemberg
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Waldkliniken Eisenberg, Eisenberg, Thuringia
- Nottingham University Hospital NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No